CLINICAL TRIAL: NCT00841451
Title: Pulmonary Vein Isolation Outcomes With Eicosapentaenoic Acid (EPA)and Docosahexaenoic Acid (DHA)
Brief Title: Pulmonary Vein Isolation Outcomes With Fish Oils
Acronym: PUFA
Status: No longer available | Type: Expanded Access
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-123
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Persistent; Paroxysmal; Pulmonary Vein isolation; Omega three fatty acids; Fish Oils
MeSH Terms: conditions — Atrial Fibrillation | interventions — Omacor; Fish Oils

INTERVENTIONS:
Drug: Lovaza (Fish Oils) — Double blinded placebo controlled
  Other Names: Lovaza NDA021654; Omacor NDA021853

SUMMARY:
Fish oil therapy may decrease the incidence of cardiac arrhythmias. This study will test whether pre-treatment with fish oils before catheter ablation of atrial fibrillation decreases the early post operative occurrence of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal Atrial fibrillation (PAF).
* Persistent atrial fibrillation. Persistent AF is not self-limited.

Exclusion Criteria:

* Previous pulmonary vein isolation ablation procedure
* Contraindication for anticoagulation
* Permanent AF
* Severe valvular pathology
* Concurrent use of antiarrhythmic medications
* Inability to give consent
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (3):
- United States (3):
  - The Valley Hospital, Ridgewood, New Jersey
  - University Medical Practice Associates 425 West 59th St. #9C, New York, New York
  - St.Luke's Hospital 1111 Amsterdam Ave. 3rd Floor Cardiology, New York, New York